CLINICAL TRIAL: NCT03274245
Title: Implementing and Evaluating a Multi-Level Intervention to Increase Latrine Use and Safe Feces Disposal Among Latrine Owning Households in Rural Puri District, Odisha, India
Brief Title: Evaluating a Latrine Use Intervention in Odisha, India
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Bethany Caruso, Post Doctoral Fellow, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB00098293
Record Dates: First submitted 2017-09-05; First posted 2017-09-06 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Latrine Usage
Keywords: Public Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Latrine Use (Experimental): Men and women in villages randomized to the latrine use arm will receive the intervention package that includes activities at the community and household levels, with additional activities and hardware for mothers of children under five.
  Interventions: Behavioral: Intervention Package
- Control Group (No Intervention): Men and women in villages randomized to the control group will not receive an intervention.
- Qualitative Research Group (Experimental): Six villages unassociated with the randomized villages will engage in qualitative research. Three villages will receive the intervention. Three villages will not receive the intervention.
  Interventions: Behavioral: Intervention Package; Other: Qualitative Research

INTERVENTIONS:
Behavioral: Intervention Package — * Community Level:
    * Palla: songs and skits to increase knowledge of and motivation for latrine use, pit emptying, safe feces disposal;
    * Transect Walk: village walk to identify and mark feces in community;
    * Community meetings: sex-segregated meetings with village members to decide on an action plan to increase community cleanliness/reduce open defecation;
    * Wall painting: village map noting households that use latrines always.
  * Sub-Community level:
    * Mothers meeting: For caregivers with children under age 5, to provide knowledge of and hardware for safe child feces disposal.
  * Household Level:
    * Household visits: to those with latrines to motivate use;
    * Latrine repairs: for households with non-functional latrines to make functional.
  Arms: Latrine Use; Qualitative Research Group
Other: Qualitative Research — For villages receiving the intervention package, investigators will engage community members through qualitative interviews to gain their perception of the intervention, what they thought of the intervention activities, what information they recall, what aspects they enjoyed or disliked, if they had barriers to attendance or participation.
  For the three villages not receiving the intervention, investigators will conduct qualitative interviews to determine additional barriers and determinants of latrine use to identify other potential intervention strategies.
  Arms: Qualitative Research Group

SUMMARY:
The objective of this research is to evaluate an intervention focused on increasing latrine use in rural Odisha India. The present study builds off of previous research, which resulted in the design of an intervention to increase latrine use. This research evaluates the intervention designed to determine if significant increases in latrine use are observed among those who received the intervention compared to those that did not. Qualitative research will supplement trial data collection to help explain findings and understand perceptions of the intervention.

DETAILED DESCRIPTION:
The objective of this research is to evaluate an intervention focused on increasing latrine use in rural Odisha India. The present study builds off of previous research, which resulted in the design of an intervention to increase latrine use. This research evaluates the intervention designed to determine if significant increases in latrine use are observed among those who received the intervention compared to those that did not. Qualitative research will supplement trial data collection to help explain findings and understand perceptions of the intervention.

For trial data collection, household members will be engaged in a survey that asks questions about the household, the latrine use practices of their family members, and may include additional questions about social norms attitudes, and other factors influencing latrine use.

Investigators will carry out two discrete qualitative research activities both digitally recorded: in depth interviews (IDIs) and focus group discussions (FGDs). Topics to be covered during the qualitative research include: perceptions of the intervention, reasons for using/not using latrines, motivations for sanitation behaviors.

The primary objective of the study is to evaluate a multi-level, theoretically informed intervention designed to increase latrine use for defecation among all members of households that currently own a latrine.

ELIGIBILITY:
Villages located in rural Puri district, Odisha India

Inclusion Criteria:

* Estimated 60% latrine coverage or higher
* At least 75 households
* Have a village leader willing to participate

Exclusion Criteria:

* Considered open-defecation free (ODF)
* Participants under the age of 18 will not be targeted for research-related activities, like interviews and discussions, though we will ask caregivers or other household members to provide in information about the sanitation-related behaviors of children under age 18.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11722 (Actual)
Dates: Start 2018-01-30 (Actual); Primary Completion 2019-02-18 (Actual); Study Completion 2019-04-13 (Actual)

PRIMARY OUTCOMES:
Change in Latrine Usage Rate | Baseline, Post-Intervention (Up to 1 Year)
  Latrine usage will be assessed via in-depth interviews conducted between the study team and participants. Responses to interview questions will be aggregated and categorized by common themes, and analyzed qualitatively.

SECONDARY OUTCOMES:
Change in Number of Toilets | Baseline, Post-Intervention (Up to 1 Year)
  The number of toilets in the community/village will be collected at baseline and post-intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Bethany Caruso, PhD, Principal Investigator — Emory University
Locations (1):
- Xavier Institute of Management, Bhubaneswar, Odisha, India

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Derived] Caruso BA, Sclar GD, Routray P, Nagel CL, Majorin F, Sola S, Koehne WJ 3rd, Clasen T. Effect of a low-cost, behaviour-change intervention on latrine use and safe disposal of child faeces in rural Odisha, India: a cluster-randomised controlled trial. Lancet Planet Health. 2022 Feb;6(2):e110-e121. doi: 10.1016/S2542-5196(21)00324-7. PMID 35150621
- [Derived] Caruso BA, Sclar GD, Routray P, Majorin F, Nagel C, Clasen T. A cluster-randomized multi-level intervention to increase latrine use and safe disposal of child feces in rural Odisha, India: the Sundara Grama research protocol. BMC Public Health. 2019 Mar 18;19(1):322. doi: 10.1186/s12889-019-6601-z. PMID 30885158